CLINICAL TRIAL: NCT01372202
Title: A Phase 2 Study of Paclitaxel With Cisplatin Versus Fluoropyrimidine With a Platinum Agent for Neoadjuvant Therapy in Operable Esophageal Cancer Based on CHFR Methylation Status in Diagnostic Biopsies
Brief Title: CHFR Methylation Status Esophageal Cancer Study
Acronym: J10130
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to early stopping rule
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J10130; NA_00042668 (Other: JHMIRB); R33CA127055 (NIH)
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Esophageal Cancer
Keywords: Operable; Based on CHFR Methylation Status; Diagnostic Biopsies
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Cisplatin; Oxaliplatin; Fluorouracil; Radiotherapy; Esophagectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Paclitaxel with Cisplatin along with Radiotherapy and followed by Esophagectomy
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy; Procedure: Esophagectomy
- Arm B (Active Comparator): Cisplatin or Oxaliplatin with 5-Fluorouracil along with Radiotherapy and followed by Esophagectomy
  Interventions: Drug: Cisplatin; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Radiation: Radiotherapy; Procedure: Esophagectomy
- Arm C (Active Comparator): Cisplatin with 5-Fluorouracil along with Radiotherapy and followed by Esophagectomy
  Interventions: Drug: Cisplatin; Drug: 5-Fluorouracil; Radiation: Radiotherapy; Procedure: Esophagectomy

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  Other Names: Abraxane; Taxol
  Arms: Arm A
Drug: Cisplatin — Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
  Other Names: Platinol
Drug: Oxaliplatin — Oxaliplatin 85 mg/m2 days 1, 15, 29.
  Other Names: Eloxatin
  Arms: Arm B
Drug: 5-Fluorouracil — Oxaliplatin and 5-fluorouracil:
  * Oxaliplatin 85 mg/m2 days 1, 15, 29.
  * 5-Fluorouracil 180 mg/m2 prolonged infusion starting day 1 of radiation and completing on the final day of radiation (up to 40 days)
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1-4 and 29-32.
  * Cisplatin 75 mg/m² days 1, 29.
  Other Names: 5-FU; Adrucil; Carac; Efudex; Fluorouracil
  Arms: Arm B; Arm C
Radiation: Radiotherapy — Patients will be treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
  Other Names: IMRT
Procedure: Esophagectomy — The type of resection (Ivor-Lewis, Transhiatal, etc.) will be left to the discretion of the operating surgeon. Resection will be completed between 5 and 8 weeks starting from the completion of chemotherapy and radiation (days 36 - 56).
  Other Names: Resection

SUMMARY:
This is a Phase 2 Study of Paclitaxel with Cisplatin versus Fluoropyrimidine with a Platinum Agent for Neoadjuvant Therapy in Operable Esophageal Cancer Based on CHFR Methylation Status in Diagnostic Biopsies.

DETAILED DESCRIPTION:
Primary Objectives

• To determine the rate of pathological complete response when the inclusion of paclitaxel in neoadjuvant therapy is based on the presence or absence of CHFR methylation in diagnostic biopsy specimens.

Secondary Objectives

* To determine the survival outcome with this treatment strategy.
* To determine time to disease progression with this treatment strategy.
* To determine the agreement between tumor CHFR methylation and detection in plasma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the esophagus or GE junction
2. Patient must be untreated with chemotherapy, radiation therapy, or surgery for this diagnosis of esophageal cancer. (Endoscopy with biopsy and dilation is permitted.)
3. Tumor must be located between 20 cm from the teeth endoscopically and 2 cm into the gastric cardia. Cervical esophageal cancers and true gastric cancers are excluded.
4. Stage T2-3/N0-3/M0 as determined by imaging studies and biopsy where appropriate. T4 disease is permitted if defined as resectable by the thoracic surgeon (involvement of the pleura, pericardium or diaphragm).
5. Patients must have had an endoscopic ultrasound
6. Patients must have had a staging PET scan
7. Age ≥ 18 and ≤ 75
8. ECOG performance status 0-1.
9. Surgically resectable tumor
10. Patients with a history of a curatively treated malignancy must be disease-free and have a survival prognosis that exceeds three years.
11. Patients must have adequate organ and marrow function as defined below:

    * absolute neutrophil count ≥ 1,000/mcL
    * platelets ≥ 100,000/mcL
    * total bilirubin ≤ 2 mg/dL
    * AST(SGOT)/ALT(SGPT) ≤ 2.5 X institutional ULN
    * creatinine < 1.5 X institutional ULN
12. Female patients must not be pregnant or breast feeding. Radiotherapy is associated with significant birth defects and/or non-viable fetus. Paclitaxel, cisplatin, oxaliplatin, and 5-fluorouracil have teratogenic potential. A negative pregnancy test is required within 14 days of treatment for all women of childbearing potential. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately.
13. Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients may not be receiving any investigational agents.
2. Incomplete healing from previous major surgery.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents they are assigned to.
4. Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's Wort; these drugs induce CYP3A and may decrease levels paclitaxel. 5-FU is a strong CYP2C9 inducer, and concomitant use with carvedilol, celecoxib, fosphenytoin, fluoxetine, phenytoin, warfarin and other CYP2C9 substrates should be used with caution.
5. Uncontrolled, inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. HIV-positive patients on combination antiretroviral therapy are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
7. Patients from whom biopsy tissue cannot be obtained for correlate study analysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Kelly, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Ronan Kelly, M.D., Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Paclitaxel with Cisplatin along with Radiotherapy and followed by Esophagectomy
  Paclitaxel: Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  Cisplatin: Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
  Radiotherapy: Patients will be treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
  Esophagectomy: The type of resection (Ivor-Lewis, Transhiatal, etc.) will be left to the discretion of the operating surgeon. Resection will be completed between 5 and 8 weeks starting from the completion of chemotherapy and radiation (days 36 - 56).
- Arm B: Oxaliplatin with 5-Fluorouracil along with Radiotherapy and followed by Esophagectomy
  Cisplatin: Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
  Oxaliplatin: Oxaliplatin 85 mg/m2 days 1, 15, 29.
  5-Fu: Oxaliplatin & 5-fu:
  * Oxaliplatin 85 mg/m2 days 1, 15, 29.
  * 5-Fu 180 mg/m2 prolonged infusion day 1 of radiation & completing on the final day of radiation
  Cisplatin/5-fluorouracil:
  * 5-Fu 1000 mg/m2 per day over 24 hours days 1-4 and 29-32.
  * Cisplatin 75 mg/m² days 1, 29.
  Radiotherapy: Treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
- Cisplatin With 5 Fu: Cisplatin with 5-Fluorouracil along with Radiotherapy and followed by Esophagectomy
Period: Overall Study
Arm/Group | Arm A | Arm B | Cisplatin With 5 Fu
Started | 13 | 9 | 9
Completed | 13 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 13 | 9 | 9 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 7 | 23
  >=65 years | 4 | 2 | 2 | 8
Age, Continuous [Mean (Full Range); unit: years] | 63 [54 to 72] | 67 [57 to 76] | 60 [47 to 73] | 62 [47 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 12 | 7 | 9 | 28
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 9 | 31

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response
Description: CHFR methylation status correlates with response to taxane containing platinum-based combination therapy and tumor response involving operable Esophageal Cancer. Perform analysis comparing detection of CHFR in tumor and plasma.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 13 | 9 | 9
Participants | 3 | 0 | 3

2. Secondary Outcome: Survival
Description: Overall survival with given treatment strategy.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Groups:
- Arm B: Cisplatin or Oxaliplatin, 5-Fluorouracil along , Radiotherapy and followed by Esophagectomy
  Cisplatin: Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hs days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
  Oxaliplatin: Oxaliplatin 85 mg/m2 days 1, 15, 29.
  5-Fluorouracil: Oxaliplatin and 5-fluorouracil:
  * Oxaliplatin 85 mg/m2 days 1, 15, 29.
  * 5-Fluorouracil 180 mg/m2 prolonged infusion starting day 1 of radiation and completing on the final day of radiation (up to 40 days)
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1-4 and 29-32.
  * Cisplatin 75 mg/m² days 1, 29.
  Radiotherapy: Patients will be treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
  Esophagectomy: The type of resection (Ivor-Lewis, Transhiatal, etc.) will be left to the discretion of the opera
- Arm C: Cisplatin with 5-Fluorouracil with Radiotherapy and followed by Esophagectomy
  Cisplatin: Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
    5-Fluorouracil: Oxaliplatin and 5-fluorouracil:
  * Oxaliplatin 85 mg/m2 days 1, 15, 29.
  * 5-Fluorouracil 180 mg/m2 prolonged infusion starting day 1 of radiation and completing on the final day of radiation (up to 40 days)
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1-4 and 29-32.
  * Cisplatin 75 mg/m² days 1, 29.
  Radiotherapy: Patients will be treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
  Esophagectomy: The type of resection (Ivor-Lewis, Transhiatal, etc.) will be left to the discretion of the operating surgeon. Resection will be completed between 5 and 8 weeks star
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 13 | 9 | 9
Participants | 6 | 5 | 6

3. Secondary Outcome: Time to Disease Progression
Description: To determine time to disease progression with this treatment strategy.
Time Frame: 3 years
Population: Study closed due to early stopping rule, therefore data was not collected to assess this outcome measure.
Groups:
- Arm B: Cisplatin: Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
  Oxaliplatin: Oxaliplatin 85 mg/m2 days 1, 15, 29.
  5-Fluorouracil: Oxaliplatin and 5-fluorouracil:
  * Oxaliplatin 85 mg/m2 days 1, 15, 29.
  * 5-Fluorouracil 180 mg/m2 prolonged infusion starting day 1 of radiation and completing on the final day of radiation (up to 40 days)
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1-4 and 29-32.
  * Cisplatin 75 mg/m² days 1, 29.
  Radiotherapy: Patients will be treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
  Esophagectomy: The type of resection (Ivor-Lewis, Transhiatal, etc.) will be left to the discretion of the opera
- Arm C: Cisplatin: Paclitaxel and cisplatin:
  * Paclitaxel 50 mg/m² (1 hr) days 1, 8, 15, 22, 29.
  * Cisplatin 30 mg/m² days 1, 8, 15, 22, 29.
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1- 4 and 29 - 32.
  * Cisplatin 75 mg/m² days 1, 29.
    5-Fluorouracil: Oxaliplatin and 5-fluorouracil:
  * Oxaliplatin 85 mg/m2 days 1, 15, 29.
  * 5-Fluorouracil 180 mg/m2 prolonged infusion starting day 1 of radiation and completing on the final day of radiation (up to 40 days)
  Cisplatin and 5-fluorouracil:
  * 5-Fluorouracil 1000 mg/m2 per day over 24 hours days 1-4 and 29-32.
  * Cisplatin 75 mg/m² days 1, 29.
  Radiotherapy: Patients will be treated 5 days/week at 1.8 Gy/day to a total dose of 45Gy.
  Esophagectomy: The type of resection (Ivor-Lewis, Transhiatal, etc.) will be left to the discretion of the operating surgeon. Resection will be completed between 5 and 8 weeks star
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Esophageal Tumor CHFR Methylation and Detection in Plasma
Description: To determine the agreement between tumor CHFR methylation and detection in plasma.
Time Frame: 3 years
Population: Study closed due to early stopping rule, therefore data was not collected to assess this outcome measure.
Arm/Group | Arm A | Arm B | Cisplatin With 5 Fu
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 7/13 | 4/9 | 3/9
Serious Adverse Events (participants affected / at risk) | 4/13 | 6/9 | 5/9
Other Adverse Events (participants affected / at risk) | 4/13 | 1/9 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=13) | Arm B (N=9) | Arm C (N=9)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dehydration (General disorders) | 0 (0) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial Fibrliation (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Failure to thrive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-responsive (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Thrombus (General disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=13) | Arm B (N=9) | Arm C (N=9)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Low Potassium (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 2 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 1 (2)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Calculi (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes